CLINICAL TRIAL: NCT06860100
Title: Dexmedetomidine and Tramadol on Perioperative Haemodynamics, Anxiety and Pain in Hemorrhoids Cases
Brief Title: The Effect of Preoperative Dexmedetomidine and Tramadol on Sedation, Pain and Haemodynamics in Haemorrhoids Patients
Status: Active, not recruiting | Type: Observational
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Arzu Esen Tekeli, Associated Professor Doctor, Yuzuncu Yil University
Other Study IDs: 19.11.2024/03
Record Dates: First submitted 2025-02-24; First posted 2025-03-05 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Analgesia; Sedation; Anxiety; Intraoperative Haemodynamics
Keywords: analgesia; sedation; perioperative anxiety; intraoperative aemodynamics
MeSH Terms: conditions — Agnosia; Anxiety Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Deksmedetomidine Group: Preoperative 1 mcg/kg dexmedetomidine iv infusion 10 minutes loading
- Tramadol Group: Preoerative 1 mg/kg tramadol iv infusion 10 min loading
- Control group: no medication before surgery

SUMMARY:
To investigate the effects of two different pharmacological agents used for analgesic and sedative purposes on perioperative anxiety and intraoperative haemodynamics in haemorrhoidectomy surgeries.

1. How are the effects of Dexmedetomidine and Tramadol on patient anxiety in the preoperative period?
2. Is there any difference in the evaluation of the efficacy of these drugs on postoperative VAS score?
3. How are the effects of the study drugs on intraoperative haemodynamic data?

DETAILED DESCRIPTION:
The study is planned as a randomised double blind study. The groups will be randomised and divided into two groups by closed envelope method. The person administering the drug and the person who will evaluate the patient will be different and the person making the evaluation will be unaware of which drug is administered to which patient. Preoperative evaluation of the patients included in the study will be performed at least one day before in the Anaesthesiology and Reanimation Polyclinic. Patients between 20-60 years of age, ASA I-II class, who are planned for elective haemorrhoidectomy and whose written and verbal consent is obtained will be included in the study.

Patients who are scheduled for surgery for haemorrhoids and undergo spinal anaesthesia will be included in the case group. However, patients younger than 20 years or older than 60 years, those whose consent could not be obtained, patients with severe renal and hepatic diseases, pregnant women, patients with known allergic response to the agents used and patients with coagulopathy will not be included in the study.

The study is planned as a randomised double blind study. Groups will be randomised by closed envelope method and patients will be divided into 3 groups. The people who administer the drug and the people who evaluate the patient will be different and the evaluator will be unaware of which drug is administered. Preoperative evaluation of the patients included in the study will be performed at least one day before in the Anaesthesiology and Reanimation Polyclinic. A total of 90 patients aged 20-60 years, ASA I-II class, who were planned for elective haemorrhoidectomy and whose written and verbal consent was obtained, will be included in the study.

Patients scheduled for surgery for haemorrhoids and under spinal anaesthesia will be included in the case group. However, patients younger than 20 years or older than 60 years, those whose consent could not be obtained, patients with severe renal and hepatic diseases, pregnant women, patients with known allergic response to the agents used and patients with coagulopathy will not be included in the study.

1. Group C: No drug administration before surgery (30 patients)
2. Group D: Preoperative Dexmedetomidine group (30 patients)
3. Group T: Preoperative Tramadol group (30 patients) STAI anxiety scale, VAS score and pain assessment will be applied to all groups in the preoperative evaluation room.

1-Group C-(Control group): no preoperative drug administration 2-Group D-(Dexmedetomidine group): 1 mcg/kg dexmedetomidine iv infusion 10 minutes loading 3-Group T-(Tramadol group): 1 mg/kg tramadol iv infusion 10 minutes loading All of the groups will undergo subarachnoid saddle block with 1 cc 0.5% bupivacaine heavy in the L4-L5 interval.

Intraoperative haemodynamic parameters (noninvasive blood pressure, SpO2 and heart rate) and sedation requirement will be recorded. For sedation, 1 mg midazolam will be administered intravenously to all groups. Patients will be excluded from the study if the total intraoperative sedation dose exceeds 5 mg. All data will be collected and statistically analysed and the results obtained will be interpreted.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II
* 20-60 years
* haemorrhoidectomy to be performed
* written Consent

Exclusion Criteria:

* ASA III and above Under 20 years old - over 60 years old,
* those who cannot be taken written consent
* severe renal and hepatic disease,
* pregnants,
* those with a known allergic response to the agents used
* patients with coagulopathy

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Elective haemorrhoidectomy surgery
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2025-11-17 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
STAI | Preoperative
  Preoperative STAI scores will be looked
VAS | Preoperative
  Preoperative VAS scores will be recorded

SECONDARY OUTCOMES:
haemodynamics | 5 minutes interval
  İntroperative non invasive blood pressure,

CONTACTS AND LOCATIONS:
Locations (1):
- Van Yuzuncu Yil University School of Medicine Department of Anesthesiology and Reanimation, Van, Tuşba, Turkey (Türkiye)